CLINICAL TRIAL: NCT03393858
Title: A Prospective Study of Combination of Anti-PD-1 Plus Autologous DC-CIK Cell Immunotherapy and Hyperthermia for Patients With Advanced Malignant Mesothelioma
Brief Title: Combination of Immunotherapy and Hyperthermia in Advanced Malignant Mesothelioma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The number of enrolled cases is insufficient
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jun Ren MD, PhD, Director,Capital Medical University (CMU)Cancer Center, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RF8-MM
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Cancer; Mesothelioma, Malignant
MeSH Terms: conditions — Neoplasms; Mesothelioma, Malignant | interventions — spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy plus Hyperthermia (Experimental)
  Interventions: Drug: Anti-PD-1 antibody; Biological: DC-CIK Immunotherapy; Device: Thermotron RF-8EX

INTERVENTIONS:
Drug: Anti-PD-1 antibody — Patients will receive pembrolizumab 100mg every three weeks until disease progression, unacceptable toxicity or patient refusal.
Biological: DC-CIK Immunotherapy — Mononuclear cells were collected from 50ml peripheral blood , and cultured DC-CIK cells for 15-20 days. Cells were infused back to the patients in 3 times via intravenous infusion .Patients will received at least 2 cycles of DC-CIK Immunotherapy along with 4 dosage of anti-PD-1 antibody treatment. If the evaluation of the treatment is partial response or stable disease, additional cycles were eligible.
Device: Thermotron RF-8EX — Hyperthermia for 40 minutes, with maximum temperature setted on 42℃ ± 0.5℃ as upper limit, twice a week since the 1st week of pembrolizumab for a total of 10 times.

SUMMARY:
The purpose of this study is to investigate the clinical efficacy and toxicity of anti-PD-1 monoclonal antibody plus autologous dendritic cells-cytokine induced killer cell (DC-CIK) immunotherapy combined with hyperthermia in advanced malignant mesothelioma patients.Furthermore,to characterize response to therapy,the investigators intent to explore the predictive biomarker for this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed malignant mesothelioma.
* Patients who have refused a first line platinum-based chemotherapy, or patients in progression of disease after a maximum of one line of platinum-based therapy for advanced disease.
* Estimated life expectancy > 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2.
* Age 18 to 80.
* Patients whose most recent major surgery or drug or radiation therapy for malignant tumors, if any, was at least 4 weeks ago at the subject enrollment.
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Adequate hematologic function, with WBC ≥ 3000/microliter, hemoglobin ≥ 9 g/dL (it is acceptable to have had prior transfusion), platelets ≥ 75,000/microliter; PT-INR <1.5 (unless patient is receiving warfarin in which case PT-INR must be <3), PTT <1.5X ULN Adequate renal and hepatic function, with serum creatinine < 1.5 mg/dL, bilirubin < 1.5 mg/dL (except for Gilbert's syndrome which will allow bilirubin ≤ 2.0 mg/dL), ALT and AST ≤ 2.5 x upper limit of normal.

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 6 weeks.
* Patients with a history of autoimmune disease, such as but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis,scleroderma, or multiple sclerosis. Autoimmune related thyroid disease and vitiligo are permitted.
* Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Patients with serious intercurrent chronic or acute illness, such as cardiac disease (NYHA class III or IV), hepatic disease, or other illness considered by the Principal Investigator as unwarranted high risk for investigational drug treatment.
* Patients with a medical or psychological impediment to probable compliance with the protocol should be excluded.
* Presence of an active acute or chronic infection including: a urinary tract infection, HIV (as determined by ELISA and confirmed by Western Blot). Patients with HIV are excluded based on immuno-suppression, which may render them unable to respond to the vaccine;patients with chronic hepatitis are excluded because of concern that hepatitis could be exacerbated by the injections.
* Patients on chronic steroid therapy (or other immuno-suppressives, such as azathioprine or cyclosporin A) are excluded on the basis of potential immune suppression. Patients must have had 6 weeks of discontinuation of any steroid therapy (except that used as pre-medication for chemotherapy or contrast-enhanced studies or for acute treatment (<5 days) of intercurrent medical condition such as a gout flare) prior to enrollment.
* Pregnant and nursing women should be excluded from the protocol since this research may have unknown and harmful effects on an unborn child or on young children. If the patient is sexually active, the patient must agree to use a medically acceptable form of birth control while receiving treatment and for a period of 4 months following the last therapy. It is not known whether the treatment used in this study could affect the sperm and could potentially harm a child that may be fathered while on this study.
* Patients evidence of interstitial lung disease will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival of the participants(PFS) | 24 months
  From starting date of anti-PD-1 antibody treatment until date of until the date of first documented disease progression or date of death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall survival of the participants(OS) | 24 months
  From starting date of anti-PD-1 antibody treatment until date of death from any cause.
Assessment of Patient- Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | 24 months
  To assess and compare the PRO-CTCAE by patients receiving immunotherapy
Safety (adverse events) | 24 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical Unvierstiy Cancer Center/ Beijing Shijitan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No